CLINICAL TRIAL: NCT06847360
Title: Home-Based Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) for Pain and Symptom Management Among Young Adults With Irritable Bowel Syndrome (IBS)
Brief Title: Home-based Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) for IBS Pain
Acronym: IBS-taVNS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Florida State University (Other); Rutgers University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000039295; R34AT012917-01A1 (NIH)
Record Dates: First submitted 2025-01-29; First posted 2025-02-26 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Pain, Chronic; Irritable Bowel Syndrome; Symptom Cluster
MeSH Terms: conditions — Chronic Pain; Irritable Bowel Syndrome; Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding procedures will be implemented for the participants, data collectors, and data analysts to minimize bias and increase study validity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active taVNS intervention (Experimental): Active taVNS twice daily, 30 minutes per session, over 6 weeks.
  Interventions: Device: Home-based taVNS intervention
- Sham taVNS (Sham Comparator): Sham taVNS twice daily, 30 minutes per session, over 6 weeks.
  Interventions: Device: Home-based taVNS intervention

INTERVENTIONS:
Device: Home-based taVNS intervention — Home-based taVNS intervention will be administered using the non-invasive taVNS device, Parasym system (Parasym Health, Inc, London, UK).

SUMMARY:
The goal of this clinical trial is to learn the feasibility and safety of using home-based taVNS in young adults with IBS to manage their IBS-related pain and symptoms. It will also learn about participants' experience in using the home-based taVNS intervention. The main questions it aims to answer are:

* Is it feasible to use a home-based taVNS intervention for pain and symptom management among YAs with IBS?
* Is it safe and reported satisfactory to use a home-based taVNS intervention for pain and symptom management among YAs with IBS? Researchers will compare Active to Sham taVNS (a look-alike intervention that contains minimal stimulation) to see if Active taVNS works on managing IBS-related pain and symptoms.

Participants will:

* Take Active or Sham taVNS intervention for a 6-week treatment (twice daily, 30 minutes per session)
* Visit the research lab at the initial setup and the end of the 6-week treatment for checkups and tests
* Keep a diary of their symptoms and the number of times they use the taVNS.

DETAILED DESCRIPTION:
This pilot randomized controlled study aims to evaluate the feasibility, acceptability, adherence, safety, and potential implementation barriers of home-based taVNS intervention in YAs (18-29 years old) diagnosed with IBS. A two-site, two-arm, parallel, proof-of-concept randomized trial will be conducted to assess the feasibility of using the Active taVNS intervention compared with Sham taVNS in managing IBS-related pain and symptoms. Eighty YAs meeting the Rome IV diagnostic criteria of IBS will be recruited and receive either Active or Sham taVNS for pain and symptom management, along with self-management education and their usual treatment and care. After enrollment and a 2-week baseline run-in period, participants will be randomized to the Active or Sham taVNS with a 6-week treatment (30 minutes per session, twice daily for 6 weeks) and be followed up for another 6 weeks of post-treatment. Investigators will assess feasibility through recruitment rates, adherence, factors influencing adherence, safety, satisfaction, and collection of patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 29 years of age;
* Men and women;
* Diagnosis of IBS from a healthcare provider with current report of pain (volunteers asked to bring provider-verification of IBS diagnosis based on Rome IV criteria to initial study appointment);
* Experiencing moderate pain (≥3 out of 10 on numeric rating scale [NRS]) at least 4 days of the week and lasting previous three months;
* Daily access to a computer connected to the internet; and
* Able to read and speak English.

Exclusion Criteria:

* Other chronic pain condition;
* Celiac disease or inflammatory bowel disease;
* Diabetes mellitus;
* severe psychiatric condition requiring inpatient treatment in previous 6 months;
* Pregnancy or lactation;
* Regular use of opioids or other illicit substances;
* use of probiotics or antibiotics within 2 weeks from enrollment; and
* any other conditions/contraindications that prohibit the application of taVNS including but not limited to any current or past history of cardiovascular disorders, recent ear trauma, and metal implants above the level of the neck.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing taVNS - Retention rates | Baseline, week 6, week 12
  Feasibility will be assessed by evaluating the retention rate of participants who complete the taVNS sessions at 6 weeks and the follow-up at week 12. Retention rates will be calculated by comparing the number of participants who complete these timepoints with the baseline data.
Adherence of implementing taVNS - Duration of usage | week 6
  Adherence will be measured using participant self-report data and the data from the taVNS monitoring system. Actual usage time (minutes) will be extracted from the Parasym system recorder to monitor the adherence to the study protocol.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Baseline, week 6, week 12
  Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) in using the taVNS will be measured using self-reported data, including online self-monitoring diary, weekly meetings with the research team, surveys, and focus group interviews. Adverse events (AEs) will be monitored daily using the online diary with a preset form, including a 10-item survey to assess daily AEs of taVNS on 0-10 Likert scales.
Satisfaction in implementing taVNS | Baseline, week 6, week 12
  Satisfaction in using the taVNS will be measured using self-reported data including online self-monitoring diary, weekly meetings with the research team, surveys, and focus group interviews.
Change in pain intensity assessed using the Brief Pain Inventory (BPI) | Baseline, week 6 and week 12
  The BPI has a total score range of 0-10 where: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain. Total pain severity score can be found by averaging all items.
Changes in IBS symptoms using IBS Symptom Severity Scale (IBS-SSS) | Baseline, week 6, week 12
  IBS Symptom Severity Scale (IBS-SSS) will be used to measure IBS symptom severity using 100-point scales on five items: severity of abdominal pain, frequency of abdominal pain, severity of abdominal distension, dissatisfaction with bowel habits, and interference with quality of life.
Changes in IBS-related Psychophysiological Symptoms - Anxiety using Patient-Reported Outcomes Measurement Information System (PROMIS®) Anxiety 4a | Baseline, week 6, week 12
  IBS-related Psychophysiological Symptoms - Anxiety will be measured using Patient-Reported Outcomes Measurement Information System (PROMIS®) Anxiety 4a measuring for Anxiety. Raw scores range from 4 to 20, with T-scores ranging from 40.3±6.1 to 81.6±3.7. A higher PROMIS T-score represents more of the concept being measured.
Changes in IBS-related Psychophysiological Symptoms - Fatigue using Patient-Reported Outcomes Measurement Information System (PROMIS®) Fatigue 4a | Baseline, week 6, week 12
  IBS-related Psychophysiological Symptoms will be measured using Patient-Reported Outcomes Measurement Information System (PROMIS®) Fatigue 4a measuring for Fatigue. Raw scores range from 4 to 20, with T-scores ranging from 33.7±4.9 to 75.8±3.9. A higher PROMIS T-score represents more of the concept being measured.
Changes in IBS-related Psychophysiological Symptoms - Depression using Patient-Reported Outcomes Measurement Information System (PROMIS®) Depression 4a | Baseline, week 6, week 12
  IBS-related Psychophysiological Symptoms will be measured using Patient-Reported Outcomes Measurement Information System (PROMIS®) measuring for Depression. Raw scores range from 4 to 20, with T-scores ranging from 41.0±6.2 to 70.4±2.6. A higher PROMIS T-score represents more of the concept being measured.
Changes in IBS-related Psychophysiological Symptoms - Applied Cognition using Patient-Reported Outcomes Measurement Information System (PROMIS®) Applied Cognition Abilities 4a | Baseline, week 6, week 12
  IBS-related Psychophysiological Symptoms will be measured using Patient-Reported Outcomes Measurement Information System (PROMIS®) measuring for Applied Cognition. Raw scores range from 4 to 20, with T-scores ranging from 30.1± 4.44 to 63.8±5.2. A higher PROMIS T-score represents more of the concept being measured.
Changes in IBS-related Psychophysiological Symptoms - Sleep using Patient-Reported Outcomes Measurement Information System (PROMIS®) Sleep Disturbance 4a | Baseline, week 6, week 12
  IBS-related Psychophysiological Symptoms will be measured using Patient-Reported Outcomes Measurement Information System (PROMIS®) Sleep Disturbance 4a measuring for sleep disturbance. Raw scores range from 4 to 20, with T-scores ranging from 32.0±5.2 to 73.3±4.6. A higher PROMIS T-score represents more of the concept being measured.
Changes in IBS related psychosocial factors - Stress using Perceived Stress Scale-10 (PSS-10) | Baseline, week 6, week 12
  IBS related psychosocial factors - stress will be measured using Perceived Stress Scale-10 (PSS-10). The scale consists of 10 items each rated on a 5-point rating scale from "never" to "very often." The sum score ranges from 0 to 40, where a higher score indicates a higher level of stress.
Changes in IBS-related quality of life using IBS-Quality of Life (IBS-QOL) Questionnaire | Baseline, week 6, week 12
  IBS-related quality of life will be measured using IBS-Quality of Life (IBS-QOL) Questionnaire. The IBS-QOL consists of 34 self-report items and a five-point Likert scale (0 to 4) is used to measure participants' feelings. The total scores are calculated as the sum of all item scores ranging from 0 to 136 and higher scores show better QOL.
Changes in IBS related psychosocial factors - Self-Efficacy using IBS Self-Efficacy Scale (IBS-SE) | Baseline, week 6, week 12
  IBS Self-Efficacy Scale (IBS-SE) will be used to measure patients' confidence in their ability to manage IBS abdominal pain and episodes using a 7-point Likert scale on 25 items. The sum of the items derives a total score ranging from 25 to 175. Higher scores indicate higher levels of self-efficacy for IBS symptom control and management.
Changes in IBS related psychosocial factors - Pain Catastrophizing using Brief Pain Catastrophizing Scale (Brief-PCS) | Baseline, week 6, week 12
  Brief Pain Catastrophizing Scale (Brief-PCS) will be used to measure the perception of pain catastrophizing, which includes 4-item brief version of the PCS, using 5-point scale. The Brief-PCS has a score range 0-16 and higher scores indicate a higher level of catastrophizing.
Changes in IBS related psychosocial factors - Coping using Coping Strategies Questionnaire-Revised (CSQ-R) | Baseline, week 6, week 12
  Coping Strategies Questionnaire-Revised (CSQ-R) will be used to measure coping strategies in managing IBS-related pain. It is a 27-item questionnaire designed to assess six cognitive coping responses to pain. Subjects rate the frequency of using each coping strategy and perceived control over their pain on a 7-point Likert-type scale (0-6). Total scores range from 0 to 162 with higher scores indicating greater use of coping strategies.
Changes in IBS related psychosocial factors - Emotion Regulation using Difficulties in Emotion Regulation Scale (DERS) | Baseline, week 6, week 12
  Difficulties in Emotion Regulation Scale (DERS) will be used to measure IBS related emotion regulation. DERS is a 36-itme self-report measure of individuals' abilities to respond to emotional experience in a goal-oriented manner, using a 5-point Likert scale. Total scores range from 36 to 180, with higher scores indicating greater difficulties in emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei S Cong, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Scientific data will be shared as soon as possible. Scientific data included in published manuscripts will be available at the time of publication; all other generated scientific data will be shared no later than the end of the award period. Under the current repository policies, data published in Dryad are permanently archived and available for broader research.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Scientific data will be shared as soon as possible. Scientific data included in published manuscripts will be available at the time of publication; all other generated scientific data will be shared no later than the end of the award period. Under the current repository policies, data published in Dryad are permanently archived and available for broader research.
Access Criteria: By the request of the researchers